CLINICAL TRIAL: NCT04381728
Title: PREvention of Intrauterine Adhesion After Hysteroscopic Surgery With Novel deGradable Film
Acronym: PREG1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Womed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREG1
Record Dates: First submitted 2020-04-28; First posted 2020-05-11 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Intrauterine Adhesion
Keywords: myomectomy; Intrauterine adhesion; hysteroscopy
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Womed Leaf (Experimental): At the end of the hysteroscopic myomectomy, Womed Leaf is delivered in the uterus thanks to a 5mm diameter, flexible inserter. Then an endovaginal ultrasound will be performed to assess the positioning of the uterine film.
  Another ultrasound will be performed at 2 hours, prior to patient discharge in order to record images of the uterine film deployment.
  A second look hysteroscopy will performed at 4-8 weeks to evaluate the presence of intrauterine adhesion.
  Interventions: Device: Womed Leaf

INTERVENTIONS:
Device: Womed Leaf — Womed Leaf uterine film will be inserted immediately after the myomectomy, following per-operative hysterometry.

SUMMARY:
Intrauterine adhesions (IUA) are the major long-term complication of intrauterine procedures and are associated with pelvic pain, menstrual disorders, obstetrical complication and infertility.

Womed Leaf is a medical device specifically designed for intrauterine use that prevents intra-uterine adhesions. It is a film that acts as a mechanical barrier to keep uterus walls separated during healing. It is then naturally discharged through the cervix and vagina in less than 30 days.

The PREG1 clinical investigation is designed to evaluate Womed Leaf safety under clinical conditions, in women scheduled for a hysteroscopic myomectomy as well as its efficacy.

DETAILED DESCRIPTION:
Intrauterine adhesions (IUA) are defined as "fibrous strings at opposing walls of the uterus and/or cervix leading to partial or complete obliteration of the cavity". IUAs are the major long-term complication of intrauterine procedures and are associated with pelvic pain, menstrual disorders, obstetrical complications and infertility.

Womed Leaf™ is a sterile, degradable polymer film specifically design for intrauterine use. It is inserter in the uterus like an intrauterine device. Once released it will self-deploy into the uterine cavity to form a mechanical barrier keeping uterus walls separated during healing, for several days, thus preventing the formation or recurrence of intrauterine adhesions. It is degraded and discharged naturally through the cervix and vagina in less than 30 days.

The PREG1 clinical investigation is a prospective multicenter, single arm study, designed to evaluate Womed Leaf safety under clinical conditions, in women scheduled for a hysteroscopic myomectomy as well as its efficacy in preventing IUA at second look hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 40 years AND no childbearing wish, OR history of permanent sterilization;
* Subject scheduled for hysteroscopic myomectomy for one or more myoma(s) where one myoma is at least 10 mm in size (≥10mm) as estimated by pre-operative ultrasound measurement of the largest diameter,
* Hysterometry prior to device insertion ≥ 6cm and ≤ 9cm.
* Subjects who are willing to provide a written informed consent as approved by the applicable Ethics Committee prior to participating in this clinical investigation.
* Subjects who can comply with the study follow-up or other study requirements

Exclusion Criteria:

Pre-operative exclusion criteria:

* Current pregnancy
* Abnormal uterine cavity according to ESHRE classification I to VI, such as unicornis, bicornis, septate, duplex
* Known or suspected endometrial hyperplasia
* Medical history of cervical or endometrial cancer
* Active pelvic infection or medical history of pelvic peritonitis
* Intrauterine device in situ
* Known contraindication or hypersensitivity to PEO or PLA, and to medications such as aspirin….
* Concurrent medical condition with a life expectancy of less than 12 months
* Full endometrial ablation

Per-operative exclusion criteria:

* Adenomyosis
* Inflammation (endometritis)
* Abnormal uterine cavity
* Hysterometry < 6cm or >9cm
* Any complication during the intervention that is deemed to potentially interfere with the objective of the study by the investigator

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- UZ Gent, Ghent, Belgium
- France (2):
  - CHU Nîmes, Nîmes
  - CHU Bicêtre (APHP), Paris
- Netherlands (3):
  - Bergman Clinics, Amsterdam
  - Zaans Medical Center, Amsterdam
  - Isala Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participant data is planed

REFERENCES:
- [Derived] Weyers S, Capmas P, Huberlant S, Dijkstra JR, Hooker AB, Hamerlynck T, Debras E, De Tayrac R, Thurkow AL, Fernandez H. Safety and Efficacy of a Novel Barrier Film to Prevent Intrauterine Adhesion Formation after Hysteroscopic Myomectomy: The PREG1 Clinical Trial. J Minim Invasive Gynecol. 2022 Jan;29(1):151-157. doi: 10.1016/j.jmig.2021.07.017. Epub 2021 Jul 31. PMID 34343712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six centers in France, Belgium and the Netherlands participated in the trial. Between November 2019 and January 2021, 23 patients were enrolled into the study.
Groups:
- Womed Leaf: At the end of the hysteroscopic myomectomy, Womed Leaf was delivered in the uterus thanks to a 5mm diameter, flexible inserter. Then an endovaginal ultrasound was performed to assess the positioning of the uterine film.
  Another ultrasound was performed at 2 hours, prior to patient discharge in order to record images of the uterine film deployment.
  A second look hysteroscopy was performed at 4-8 weeks to evaluate the presence of intrauterine adhesion.
Period: Overall Study
Arm/Group | Womed Leaf
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 7
  Belgium | 4
  France | 12
Myoma type (FIGO classification) [Count of Participants; unit: Participants]
  FIGO type 0 (pedunculated intracavitary) | 4
  FIGO type 1 (< 50% intramural) | 10
  FIGO type 2 (> 50% intramural) | 9
Mean number of tumor resected [Mean (Standard Deviation); unit: tumors resected] | 1.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Safety (Adverse Events)
Description: The number and severity of polymer film related adverse event
Time Frame: 30 days
Measure: Number; unit: device related adverse event
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
device related adverse event | 0

2. Primary Outcome: Efficacy (Rate of Patient With no IUA)
Description: Freedom from intrauterine adhesion
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
Participants | 20

3. Primary Outcome: Efficacy (Intrauterine Adhesion Severity According to AFS Classification)
Description: Severity of IUAs according to American Fertility Society (AFS) classification systems of adhesions.
  Pronostic classification => Hysteroscopy score Stade I (mild) => 1-4 Stade II (moderate) => 5-8 Stade III (severe) => 9-12
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
Participants
  mild adhesions | 2
  moderate adhesions | 1

4. Primary Outcome: Efficacy (Intrauterine Adhesion Severity According to ESGE Classification)
Description: Severity of IUAs according to European Society of Gynecological Endoscopy (ESGE) classification systems of adhesions.
  I => Thin or filmy IUA easily ruptured by HSC sheath alone. Cornual areas normal II => Singular dense IUA connecting separate parts of the uterine cavity. Visualization of both tubal ostia possible. Cannot be ruptured by HSC sheath alone IIa => Occluding IUA only in the region of the internal cervical os. Upper uterine cavity normal III => Multiple dense IUA connecting separate parts of the uterine cavity. Unilateral obliteration of ostial areas of the tubes IV => Extensive dense IUA with (partial) occlusion of the uterine cavity. Both tubal ostial areas (partially) occluded Va => Extensive endometrial scarring and fibrosis in combination with grade I or grade II IUA with amenorrhea or pronounced hypomenorrhea Vb => Extensive endometrial scarring and fibrosis in combination with grade III or grade IV IUA with amenorrhea
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
Participants
  Grade II | 1
  Grade III | 2

5. Secondary Outcome: Adverse Events
Description: Number of adverse events (AE) at 30 days
Time Frame: 30 days
Measure: Number; unit: adverse events
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
adverse events | 3

6. Secondary Outcome: Device Technical Success
Description: Defined as the rate of success of the following 2 steps : insertion and release
Time Frame: During operation: T=0
Measure: Count of Participants; unit: Participants
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
Participants | 23

7. Secondary Outcome: Womed Leaf Residuals
Description: Presence of Womed Leaf residuals in the uterus
Time Frame: At second look hysteroscopy: 4-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
Participants | 0

8. Secondary Outcome: Womed Leaf Discharge Feedback : Time Interval in Days Between Surgery and Discharge
Description: Uterine film discharge experience as recalled by subject using a survey to be asked to the patient
Time Frame: At second look hysteroscopy: 4-8 weeks
Population: 10 patients did not notice the discharge of the device
Measure: Median (Full Range); unit: days
Arm/Group | Womed Leaf
Number analyzed (Participants) | 13
days | 6 [1 to 15]

9. Secondary Outcome: Device Manipulation
Description: Device manipulation duration from insertion to withdrawal.
Time Frame: During intervention: T=0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Womed Leaf
Number analyzed (Participants) | 23
minutes | 2 (0)

10. Secondary Outcome: Womed Leaf Discharge Feedback Questionnaire (Polymer Tolerance Assessed on a Scale From 1 (no Discomfort) to 10 (Extremely Disturbing))
Description: Uterine film discharge experience as recalled by subject using a survey to be asked to the patient
Time Frame: At second look hysteroscopy: 4-8 weeks
Population: 10 patients did not notice the discharge of the device
Measure: Mean (Standard Deviation); unit: scale from 1 (no discomfort) to 10
Arm/Group | Womed Leaf
Number analyzed (Participants) | 13
scale from 1 (no discomfort) to 10 | 1.9 (1.8)

ADVERSE EVENTS:
Time Frame: 30 days after hysteroscopic myomectomy and device insertion
Arm/Group | Womed Leaf
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Womed Leaf (N=23)
Bleeding (Surgical and medical procedures) | 1
renal colic (General disorders) | 1
Hematoma (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04381728/Prot_000.pdf